CLINICAL TRIAL: NCT02530957
Title: Comparison of Two Methods of Preoxygenation Before Oro Tracheal Intubation in the Hypoxemic Patient in Intensive Care Unit : Non Invasive Ventilation (NIV) + High Flow Nasal Cannula Oxygen Versus NIV Alone : a Randomized Controlled Study
Brief Title: Non Invasive Ventilation Combined to High Flow Nasal Cannula Oxygen for Preoxygenation of Hypoxemic ICU Patients
Acronym: OPTINIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 9543; 2015-A00708-41 (Other: RCB number)
Record Dates: First submitted 2015-08-07; First posted 2015-08-21 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Intubation Intraesophageal
Keywords: Intubation; Preoxygenation; Complications; Non invasive ventilation; High flow nasal cannula
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventional (Experimental): In the interventional group, a preoxygenation by NIV (PS of 10 cm H2O, PEEP of 5 cm H2O, FiO2 = 100%) combined to HNFC (Flow of 60L/min, FiO2 = 100%) is applied.
  Interventions: Device: Non invasive ventilation + High flow nasal cannula oxygen
- Reference (Other): In the reference group, a preoxygenation by NIV only (PS of 10 cm H2O, PEEP of 5 cm H2O, FiO2 = 100%) is applied.
  Interventions: Device: Non invasive ventilation

INTERVENTIONS:
Device: Non invasive ventilation + High flow nasal cannula oxygen — In the interventional group, a preoxygenation by NIV (venturi mask of Intersurgical or Respironics mask) with PS of 10 cm H2O, PEEP of 5 cm H2O, FiO2 = 100% and combined to HNFC (nasal cannula oxygen of Fisher and Paykel) with Flow of 60L/min, FiO2 = 100% is applied.
  Arms: Interventional
Device: Non invasive ventilation — In the reference group, a preoxygenation by NIV (venturi mask of Intersurgical or Respironics mask) only, with PS of 10 cm H2O, PEEP of 5 cm H2O, FiO2 = 100% is applied.
  Arms: Reference

SUMMARY:
Tracheal intubation is a challenging procedure in Intensive Care Unit (ICU), associated with severe life threatening complications. To decrease these complications, preoxygenation is recommended. Non invasive ventilation (NIV) increase effectiveness of preoxygenation, applying a positive end expiratory pressure (PEEP). High-flow nasal cannula oxygen (HFNC) improves oxygenation by increasing end-expiratory lung volume and has a potential of apneic oxygenation. The association of NIV and HFNC for preoxygenation in hypoxemic ICU patients has never been evaluated. The aim of this study is to determine if HFNC combined to NIV could have therapeutic advantages over NIV alone for preoxygenation in the ICU patients intubated for hypoxemic acute respiratory failure.

DETAILED DESCRIPTION:
Patients admitted in Intensive Care Unit (ICU) often need respiratory support. Endotracheal intubation procedure in ICU is associated with severe life threatening complications. In order to decrease the incidence of complications including hypoxemia during intubation procedure, a preoxygenation is recommended, consisting in the administration of pure oxygen before intubation.

Recent data suggest that NIV use for preoxygenation of patients with acute respiratory failure is associated with less hypoxemia during intubation procedure than classic preoxygenation with facial mask. Indeed, associating Pressure Support (PS) with Positive end expiratory pressure (PEEP) limits the alveolar collapse and atelectasis formation. NIV is now used by a lot of of teams for preoxygenation of patients with acute respiratory failure in ICU.

However, although NIV is effective to reduce hypoxemia during intubation procedure, NIV mask has to be taken off after preoxygenation in order to allow the passage of the oro tracheal tube through the mouth. The hypoxemic patient does not receive oxygen during this period, which participates to the episodes of major hypoxemia during intubation.

In contrast, HFNC, which delivers high flow heated and humidified oxygen and air via nasal prongs at a prescribed fraction of inspired oxygen and a maximum flow of 60 L/min can be pursued during the intubation procedure. Some very recent studies suggest that HNFC could allow apneic oxygenation.

Although use of HFNC combined to NIV may have potential advantages over conventional NIV for preoxygenation before intubation in hypoxemic ICU patients, this technique of preoxygenation has never been assessed and benefit remains to be established.

The OPTINIV study aims to compare the effects of preoxygenation with combination of NIV and HFNC versus NIV alone on lowest oxygen saturation during intubation procedure of ICU patients intubated for acute respiratory failure.

Study design and population The OPTINIV trial is an investigator initiated multicenter randomized controlled two-arm blinded trial.

Local investigators screen consecutive patients intubated in ICU, with an acute respiratory failure (respiratory rate > 25/min) and hypoxemia. Hypoxemia is defined by the need of a fraction inspirated in oxygen (FiO2)>50% to maintain a saturation of arterial blood with oxygen as measured by pulse oximetry (SpO2)>90% and a partial pressure of oxygen in the arterial blood (PaO2)/FiO2 ratio<300 mmHg under mask oxygen therapy with a flow of 15L/min (measured during the 4 hours before inclusion).

Patients fulfilling one or more of the following criteria will not be included: nonadult patients (age <18 years), pregnant, protected persons, intubation in case of cardio circulatory arrest, nasopharyngeal obstacle contraindicating the use of HNFC.

Ethics and consent The Institutional Review Board of the University Hospital of Montpellier (France) approved the trial. By May 2015, the study had been approved by a central ethics committee (Committee for the Protection of Persons, Montpellier, France) with the registration number IDRCB 2015-A00708-41.

All patients or their next will asked for signed informed consent, as required by the institutional review board in accordance with the Declaration of Helsinki or emergency procedure allowed inclusion as a part of care in acute situation according the French Law.

Data collection The following data will be collected and registered before intubation: demographic data : age, sex, weight, height, date and hour of intubation, severity scores (Simplified Acute Physiologic Score (SAPS) II at admission, Sequential Organ Failure Assessment (SOFA) score on the day of the procedure), type of admission, reason of admission in ICU, indication of intubation, comorbidities, nature and number of operators, formation, fluid loading before intubation, arterial pressure and lowest saturation, therapeutic by vasopressor drugs or non invasive ventilation, predictive criteria of difficult intubation (including the MACOCHA score).

During the preoxygenation, will be recorded : need to change the method of preoxygenation and the reasons for changing, size of intubation tube, vital parameters : oxygen saturation at the beginning and at the end of the preoxygenation, lowest saturation, lowest and highest arterial pressure and heart rate, length and difficulty of preoxygenation.

During the intubation procedure, the following parameters will be collected : hypnotic and neuromuscular blocker used and dose, oxygen saturation at the beginning and at the end, lowest saturation, total length of intubation procedure, difficult intubation, number of operators, number of attempts, Cormack grade, traction force on the laryngoscope, Sellick manoeuver, occurrence of complications related to intubation.

After the intubation procedure (until one hour after): a thorax X-ray will be done, and arterial blood gases. Complications related to intubation will be collected.

Length of mechanical ventilation, length of stay in ICU, mortality at day 28 will be recorded.

Trial interventions Patients eligible for inclusion are randomly assigned to the interventional group or to the reference group. In the interventional group, a preoxygenation by NIV (PS of 10 cm H2O, PEEP of 5 cm H2O, FiO2 = 100%) combined to HNFC (Flow of 60L/min, FiO2 = 100%) is applied. HFNC will applied along all the intubation procedure including the apnea period. In the reference group, a preoxygenation by NIV only (PS of 10 cm H2O, PEEP of 5 cm H2O, FiO2 = 100%) will be applied.

Outcomes Primary outcome variable is the lowest oxygen saturation collected by pulse oxymetry during the intubation procedure. The intubation procedure lasts from the beginning of the first laryngoscopy to the confirmation of the orotracheal intubation.

Secondary outcome variables are preoxygenation quality, complications related to intubation (severe : severe hypoxemia defined by lowest saturation < 80 %, severe cardiovascular collapse, defined as systolic blood pressure less than 65 mm Hg recorded at least one time or less than 90 mm Hg that lasted 30 minutes despite 500-1,000 ml of fluid loading (crystalloids or colloids solutions) or requiring introduction of vasoactive support, cardiac arrest, death during intubation; moderate: difficult intubation, arrhythmias, esophageal intubations, agitation, pulmonary aspiration, dental injuries), morbidity in ICU (length of stay, length of mechanical ventilation, mortality at 28 days).

Statistical analysis Quantitative variables will be expressed as means (standard deviation) or medians (interquartiles 25%-75%) and compared using the student t test or the Wilcoxon test as appropriate (Gaussian or non Gaussian variables). Qualitative variables will be compared using the chi 2 test or the Fisher test as appropriate.

A linear regression will be used to adjust the relation of lowest oxygen saturation during intubation procedure and group of inclusion. A multivariate model will be established.

A p-value of ≤ .05 will be considered statistically significant. The statistical analysis will be performed by the medical statistical department of the Montpellier University Hospital with the help of statistical software (SAS, version 9.3; SAS Institute; Cary, NC and R, version 2.14.1).

ELIGIBILITY:
Inclusion Criteria:

* Adult hypoxemic patients
* Patients intubated in the ICU for acute respiratory failure (Hypoxemia is defined by the need of a FiO2>50% to maintain a SpO2>90% and a PaO2/FiO2 ratio<300 mmHg under mask oxygen therapy with a flow of 15L/min (measured during the 4 hours before inclusion)).

Exclusion Criteria:

* non adult patients (age <18 years)
* pregnant woman
* protected persons
* Patient intubated in case of cardio circulatory arrest
* Patient with nasopharyngeal obstacle contraindicating the use of HNFC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06-23 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2016-03-17 (Actual)

PRIMARY OUTCOMES:
Lowest oxygen saturation | 1 years

SECONDARY OUTCOMES:
Number of complications related to intubation | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Samir JABER, M.D, Ph.D, Principal Investigator — Departement of Unit Care in Montpellier
Locations (1):
- Centre Hospitalier Universitaire Montpellier, Saint Eloi, Montpellier, Languedoc-Roussillon, France

REFERENCES:
- [Background] De Jong A, Molinari N, Terzi N, Mongardon N, Arnal JM, Guitton C, Allaouchiche B, Paugam-Burtz C, Constantin JM, Lefrant JY, Leone M, Papazian L, Asehnoune K, Maziers N, Azoulay E, Pradel G, Jung B, Jaber S; AzuRea Network for the Frida-Rea Study Group. Early identification of patients at risk for difficult intubation in the intensive care unit: development and validation of the MACOCHA score in a multicenter cohort study. Am J Respir Crit Care Med. 2013 Apr 15;187(8):832-9. doi: 10.1164/rccm.201210-1851OC. PMID 23348979
- [Background] Jaber S, Amraoui J, Lefrant JY, Arich C, Cohendy R, Landreau L, Calvet Y, Capdevila X, Mahamat A, Eledjam JJ. Clinical practice and risk factors for immediate complications of endotracheal intubation in the intensive care unit: a prospective, multiple-center study. Crit Care Med. 2006 Sep;34(9):2355-61. doi: 10.1097/01.CCM.0000233879.58720.87. PMID 16850003
- [Background] De Jong A, Jung B, Jaber S. Intubation in the ICU: we could improve our practice. Crit Care. 2014 Mar 18;18(2):209. doi: 10.1186/cc13776. No abstract available. PMID 25029179
- [Background] De Jong A, Futier E, Millot A, Coisel Y, Jung B, Chanques G, Baillard C, Jaber S. How to preoxygenate in operative room: healthy subjects and situations "at risk". Ann Fr Anesth Reanim. 2014 Jul-Aug;33(7-8):457-61. doi: 10.1016/j.annfar.2014.08.001. Epub 2014 Aug 29. PMID 25168301
- [Background] Baillard C, Fosse JP, Sebbane M, Chanques G, Vincent F, Courouble P, Cohen Y, Eledjam JJ, Adnet F, Jaber S. Noninvasive ventilation improves preoxygenation before intubation of hypoxic patients. Am J Respir Crit Care Med. 2006 Jul 15;174(2):171-7. doi: 10.1164/rccm.200509-1507OC. Epub 2006 Apr 20. PMID 16627862
- [Background] Jaber S, Michelet P, Chanques G. Role of non-invasive ventilation (NIV) in the perioperative period. Best Pract Res Clin Anaesthesiol. 2010 Jun;24(2):253-65. doi: 10.1016/j.bpa.2010.02.007. PMID 20608561
- [Background] Vourc'h M, Asfar P, Volteau C, Bachoumas K, Clavieras N, Egreteau PY, Asehnoune K, Mercat A, Reignier J, Jaber S, Prat G, Roquilly A, Brule N, Villers D, Bretonniere C, Guitton C. High-flow nasal cannula oxygen during endotracheal intubation in hypoxemic patients: a randomized controlled clinical trial. Intensive Care Med. 2015 Sep;41(9):1538-48. doi: 10.1007/s00134-015-3796-z. Epub 2015 Apr 14. PMID 25869405
- [Background] Miguel-Montanes R, Hajage D, Messika J, Bertrand F, Gaudry S, Rafat C, Labbe V, Dufour N, Jean-Baptiste S, Bedet A, Dreyfuss D, Ricard JD. Use of high-flow nasal cannula oxygen therapy to prevent desaturation during tracheal intubation of intensive care patients with mild-to-moderate hypoxemia. Crit Care Med. 2015 Mar;43(3):574-83. doi: 10.1097/CCM.0000000000000743. PMID 25479117
- [Background] Chanques G, Riboulet F, Molinari N, Carr J, Jung B, Prades A, Galia F, Futier E, Constantin JM, Jaber S. Comparison of three high flow oxygen therapy delivery devices: a clinical physiological cross-over study. Minerva Anestesiol. 2013 Dec;79(12):1344-55. Epub 2013 Jul 15. PMID 23857440
- [Background] Chanques G, Jaber S. [Unexpected progress of an old intensive care therapy, oxygen: towards more comfort and less mechanical ventilation...]. Rev Mal Respir. 2013 Oct;30(8):605-8. doi: 10.1016/j.rmr.2013.07.006. Epub 2013 Aug 27. No abstract available. French. PMID 24182647
- [Background] Hedenstierna G, Rothen HU. Atelectasis formation during anesthesia: causes and measures to prevent it. J Clin Monit Comput. 2000;16(5-6):329-35. doi: 10.1023/a:1011491231934. PMID 12580216
- [Background] Hedenstierna G, Edmark L. The effects of anesthesia and muscle paralysis on the respiratory system. Intensive Care Med. 2005 Oct;31(10):1327-35. doi: 10.1007/s00134-005-2761-7. Epub 2005 Aug 16. PMID 16132894
- [Background] Kolettas A, Grosomanidis V, Kolettas V, Zarogoulidis P, Tsakiridis K, Katsikogiannis N, Tsiouda T, Kiougioumtzi I, Machairiotis N, Drylis G, Kesisis G, Beleveslis T, Zarogoulidis K. Influence of apnoeic oxygenation in respiratory and circulatory system under general anaesthesia. J Thorac Dis. 2014 Mar;6 Suppl 1(Suppl 1):S116-45. doi: 10.3978/j.issn.2072-1439.2014.01.17. PMID 24672687
- [Background] Engstrom J, Hedenstierna G, Larsson A. Pharyngeal oxygen administration increases the time to serious desaturation at intubation in acute lung injury: an experimental study. Crit Care. 2010;14(3):R93. doi: 10.1186/cc9027. Epub 2010 May 24. PMID 20497538
- [Background] Griesdale DE, Bosma TL, Kurth T, Isac G, Chittock DR. Complications of endotracheal intubation in the critically ill. Intensive Care Med. 2008 Oct;34(10):1835-42. doi: 10.1007/s00134-008-1205-6. Epub 2008 Jul 5. PMID 18604519
- [Background] Jaber S, Jung B, Corne P, Sebbane M, Muller L, Chanques G, Verzilli D, Jonquet O, Eledjam JJ, Lefrant JY. An intervention to decrease complications related to endotracheal intubation in the intensive care unit: a prospective, multiple-center study. Intensive Care Med. 2010 Feb;36(2):248-55. doi: 10.1007/s00134-009-1717-8. Epub 2009 Nov 17. PMID 19921148
- [Background] De Jong A, Clavieras N, Conseil M, Coisel Y, Moury PH, Pouzeratte Y, Cisse M, Belafia F, Jung B, Chanques G, Molinari N, Jaber S. Implementation of a combo videolaryngoscope for intubation in critically ill patients: a before-after comparative study. Intensive Care Med. 2013 Dec;39(12):2144-52. doi: 10.1007/s00134-013-3099-1. Epub 2013 Sep 18. PMID 24045887
- [Background] Jung B, Clavieras N, Nougaret S, Molinari N, Roquilly A, Cisse M, Carr J, Chanques G, Asehnoune K, Jaber S. Effects of etomidate on complications related to intubation and on mortality in septic shock patients treated with hydrocortisone: a propensity score analysis. Crit Care. 2012 Nov 21;16(6):R224. doi: 10.1186/cc11871. PMID 23171852
- [Background] Futier E, Constantin JM, Pelosi P, Chanques G, Massone A, Petit A, Kwiatkowski F, Bazin JE, Jaber S. Noninvasive ventilation and alveolar recruitment maneuver improve respiratory function during and after intubation of morbidly obese patients: a randomized controlled study. Anesthesiology. 2011 Jun;114(6):1354-63. doi: 10.1097/ALN.0b013e31821811ba. PMID 21478734
- [Background] Chanques G, Constantin JM, Sauter M, Jung B, Sebbane M, Verzilli D, Lefrant JY, Jaber S. Discomfort associated with underhumidified high-flow oxygen therapy in critically ill patients. Intensive Care Med. 2009 Jun;35(6):996-1003. doi: 10.1007/s00134-009-1456-x. Epub 2009 Mar 18. PMID 19294365
- [Background] Delay JM, Sebbane M, Jung B, Nocca D, Verzilli D, Pouzeratte Y, Kamel ME, Fabre JM, Eledjam JJ, Jaber S. The effectiveness of noninvasive positive pressure ventilation to enhance preoxygenation in morbidly obese patients: a randomized controlled study. Anesth Analg. 2008 Nov;107(5):1707-13. doi: 10.1213/ane.0b013e318183909b. PMID 18931236
- [Background] De Jong A, Molinari N, Conseil M, Coisel Y, Pouzeratte Y, Belafia F, Jung B, Chanques G, Jaber S. Video laryngoscopy versus direct laryngoscopy for orotracheal intubation in the intensive care unit: a systematic review and meta-analysis. Intensive Care Med. 2014 May;40(5):629-39. doi: 10.1007/s00134-014-3236-5. Epub 2014 Feb 21. PMID 24556912
- [Background] Jaber S, De Jong A, Castagnoli A, Futier E, Chanques G. Non-invasive ventilation after surgery. Ann Fr Anesth Reanim. 2014 Jul-Aug;33(7-8):487-91. doi: 10.1016/j.annfar.2014.07.742. Epub 2014 Aug 29. PMID 25168304
- [Background] Bourgain JL, Jaber S. [Preoxygenation: conditions of success]. Ann Fr Anesth Reanim. 2010 Mar;29(3):187-8. doi: 10.1016/j.annfar.2009.12.027. Epub 2010 Jan 27. No abstract available. French. PMID 20106629
- [Background] De Jong A, Baranwal AK, Jaber S. Predictors of difficult intubation in ICU: are children and adults alike? Intensive Care Med. 2014 Nov;40(11):1769-71. doi: 10.1007/s00134-014-3429-y. Epub 2014 Aug 28. No abstract available. PMID 25164393
- [Background] De Jong A, Jaber S. [Intubation in intensive care medicine: we could improve our practices!]. Ann Fr Anesth Reanim. 2014 May;33(5):293-4. doi: 10.1016/j.annfar.2014.03.017. Epub 2014 May 9. No abstract available. French. PMID 24814026
- [Background] Mort TC. Preoxygenation in critically ill patients requiring emergency tracheal intubation. Crit Care Med. 2005 Nov;33(11):2672-5. doi: 10.1097/01.ccm.0000187131.67594.9e. PMID 16276196
- [Background] Mort TC, Waberski BH, Clive J. Extending the preoxygenation period from 4 to 8 mins in critically ill patients undergoing emergency intubation. Crit Care Med. 2009 Jan;37(1):68-71. doi: 10.1097/CCM.0b013e318192845e. PMID 19050620
- [Derived] Jaber S, Molinari N, De Jong A. New method of preoxygenation for orotracheal intubation in patients with hypoxaemic acute respiratory failure in the intensive care unit, non-invasive ventilation combined with apnoeic oxygenation by high flow nasal oxygen: the randomised OPTINIV study protocol. BMJ Open. 2016 Aug 12;6(8):e011298. doi: 10.1136/bmjopen-2016-011298. PMID 27519921